CLINICAL TRIAL: NCT05528172
Title: A Double-Masked, Randomized, Placebo-Controlled, Parallel-Group, 12-Week Treatment and 14-week Extension, Phase 3 Study to Investigate the Safety and Efficacy of Ripasudil (K-321) Eye Drops After Cataract Surgery
Brief Title: A Study to Investigate the Safety and Efficacy of Ripasudil (K-321) Eye Drops After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-321-302
Record Dates: First submitted 2022-08-25; First posted 2022-09-06 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Corneal Edema After Cataract Surgery
MeSH Terms: interventions — K-115

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants receive K-321 ophthalmic solution Four times daily(QID) for 12 Weeks followed by a 4 week follow-up period with no treatment.
  Interventions: Drug: Ripasudil
- Group B (Experimental): Participants receive K-321 ophthalmic solution Four times daily(QID) for 12 Weeks followed by a 14 week follow-up period with no treatment.
  Interventions: Drug: Ripasudil
- Group C (Placebo Comparator): Participants will receive K-321 Placebo ophthalmic solution QID for 12 Weeks followed by a 4 week follow-up period with no treatment.
  Interventions: Drug: Placebo
- Group D (Placebo Comparator): Participants will receive K-321 Placebo ophthalmic solution QID for 12 Weeks followed by a 14 week follow-up period with no treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ripasudil — K-321 ophthalmic solution
  Other Names: K-321
  Arms: Group A; Group B
Drug: Placebo — Placebo ophthalmic solution
  Arms: Group C; Group D

SUMMARY:
The purpose of this study is to assess the safety and efficacy of K-321 in subjects after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at the screening visit (Visit 1).
* Is planning to undergo cataract surgery in the study eye and has had cataract surgery at Visit 2.
* Can understand the written informed consent, provides signed written informed consent, and agrees to comply with protocol requirements before any study-specific assessment is performed.
* Meet all other inclusion criteria outlined in clinical study protocol.

Exclusion Criteria:

* Is a female subject of childbearing potential and any of the following is true:

  1. is pregnant or lactating/breastfeeding, or
  2. has experienced menarche and is not surgically sterile, not post-menopausal (no menses for the previous 12 months), or not willing to practice an effective method of birth control during the study period as determined by the Investigator (eg, oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy).
  3. has a positive urine pregnancy test result at Visit 2 before cataract surgery.
* Had intraocular surgery (non-laser surgery) in the study eye within 6 months of Visit 1.
* Had intraocular laser surgery in the study eye within 3 months of Visit 1.
* Meet any other exclusion criteria outlined in clinical study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Central Corneal Endothelial Cell Density (ECD) at Week 12 | Baseline to Week 12
  Corneal ECD measurement captured by specular microscopy

SECONDARY OUTCOMES:
Change in Central Corneal ECD | Baseline to Week 26
  Corneal ECD measurement captured by specular microscopy
Change in Peripheral Corneal ECD | Baseline to Week 26
  Corneal ECD measurement captured by specular microscopy
Change in Corneal Thickness | Baseline to Week 26
  measured in micrometers by contact ultrasound pachymetry, or optical pachymetry
Change in corneal edema | Baseline to Week 26
  assessed as either being present or absent during slit-lamp examination
Change in Best-Corrected Visual Acuity (BCVA) | Baseline to Week 26
  Measured by ETDRS scale
Change in Vision-related quality of life | Baseline to Week 26
  Visual Functioning Questionnarie-25 (VFQ 25, Version 2000)
Number of Participants with Adverse Events and Treatment Emergent Adverse Events | Baseline to Week 26
  Coded using the MedDRA dictionary (the most recent version, ver. 24.1 or later)
Safety Assessment with Slit-lamp Biomicroscopy and Dilated Fundoscopy | Baseline to Week 26
  Graded as Normal or Abnormal
Safety Assessment of Intraocular Pressure (IOP) | Baseline to Week 26
  Results will be recorded in mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Shona Pendse, MD, MMSc, Study Chair — Kowa Pharma Development Co.
Locations (45):
- United States (44):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Inland Eye Specialists, Hemet, California
  - United Medical Research Institute, Inglewood, California
  - Alvarado Eye Associates, La Mesa, California
  - SoCal Eye Physicians and Associates, Long Beach, California
  - Visionary Research Institute, Newport Beach, California
  - Pendleton Eye Center, Oceanside, California
  - North Bay Eye Associates, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Premiere Practice Management, LLC, Torrance, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Icon Eye Care, Grand Junction, Colorado
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - International Research Center, Tampa, Florida
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Durrie Vision, Overland Park, Kansas
  - Eye Care Institute/Butchertown Clinical Trials, Louisville, Kentucky
  - Maine Eye Center, Portland, Maine
  - Fraser Eye Care Center, Fraser, Michigan
  - Silverstein Eye Centers, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultantants, Ltd., St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Vance Thompson Vision-MT, Bozeman, Montana
  - Vance Thompson Vision- NE, Omaha, Nebraska
  - Wellish Vision Institute, Las Vegas, Nevada
  - Center for Sight, Las Vegas, Nevada
  - NYU Grossman School of Medicine, New York, New York
  - Seeta Eye Center, Poughkeepsie, New York
  - Vance Thompson Vision ND, West Fargo, North Dakota
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cincinnati Eye Institute, Mason, Ohio
  - Eye Care Specialists, Kingston, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Keystone Research, Austin, Texas
  - Hill Country Eye Center, Cedar Park, Texas
  - Louis M. Alpern, M.D., M.P.H.,P.A., El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Lake Travis Eye & Laser Center, Lakeway, Texas
  - DCT-Shah Research, LLC dba Discovery Clinical Trials, Mission, Texas
  - Terry Eye Associates, San Antonio, Texas
- Centro Oftalmologico Metropolitano, San Juan, Puerto Rico